CLINICAL TRIAL: NCT00627783
Title: Randomized Strategy Trial Comparing Detection of Silent Ischemia With no Detection of Silent Ischemia in Asymptomatic Patients With Type 2 Diabetes Mellitus. Effects on Cardiovascular Events.
Brief Title: Do You Need to Assess Myocardial Ischemia in Type 2 Diabetes
Acronym: DYNAMIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruiting status
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: PLATTNER, MD, HOSPICES CIVILS DE LYON
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000.217
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients are referred to a cardiologist for a systematic detection of silent ischemia by a bicycle exercise test performed according to the French Society of Cardiology protocol after washout of cardiovascular medications likely to interfere with the test. Dipyridamole Single Photon Emission Computed Tomography (SPECT) is used in patients unable to perform the exercise test, with a sub-maximal negative exercise test result or with electrocardiographic abnormalities impairing the interpretation of the exercise test. Subsequent investigations (such as coronary angiography) and treatments (such as revascularization procedures) are left at the cardiologist's decision.
  Interventions: Other: a bicycle exercise test
- Control (No Intervention): Patients are treated according current guidelines but are not referred to a cardiologist

INTERVENTIONS:
Other: a bicycle exercise test
  Arms: Intervention

SUMMARY:
DYNAMIT is a prospective, randomized, multicenter, open strategy trial run in 45 French hospitals. Diabetic patients with no evidence of coronary artery disease and at least 2 additional cardiovascular risk factors are randomized to screening for silent ischemia using a bicycle exercise test or Dipyridamole Single Photon Emission Computed Tomography (N=316), or follow-up without screening (N=315). All have access to cardiovascular prevention according current guidelines. The main end point is time to death from all causes, non-fatal myocardial infarction, non-fatal stroke, or heart failure requiring hospitalization or emergency service intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients 55 to 75 years old had type-2 diabetes and at least two of the following cardiovascular risk factors:

  * urinary albumin excretion > 30 mg/L or > 30 mg/24 hours,
  * treated or untreated hypertension,
  * treated or untreated lipid abnormality,
  * peripheral arterial disease,
  * history of transient ischemic accident,
  * tobacco consumption
  * familial history of premature cardiovascular disease.

Exclusion Criteria:

* History of myocardial infarction, coronary artery disease, or stroke,
* Previous positive stress test or myocardial perfusion imaging,
* Negative stress test or myocardial perfusion imaging within the last three years

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2000-12; Primary Completion 2005-07; Study Completion 2005-07

PRIMARY OUTCOMES:
Death from all causes, non-fatal myocardial infarction, non-fatal stroke, or heart failure requiring hospitalization or emergency service intervention, measured after a minimum follow-up of 2 years

SECONDARY OUTCOMES:
Unstable angina requiring hospitalization Coronary events Coronary revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Louis Pradel, Bron, France

REFERENCES:
- [Derived] Lievre MM, Moulin P, Thivolet C, Rodier M, Rigalleau V, Penfornis A, Pradignac A, Ovize M; DYNAMIT investigators. Detection of silent myocardial ischemia in asymptomatic patients with diabetes: results of a randomized trial and meta-analysis assessing the effectiveness of systematic screening. Trials. 2011 Jan 26;12:23. doi: 10.1186/1745-6215-12-23. PMID 21269454